

Study Title: Development and pilot evaluation of a novel cooking skills intervention to prevent

diabetes

Principal Investigator: Julia Wolfson

IRB No.: IRB00018839

PI Version Date: V2/01/05/2022

Hello. I am << Data Collector Name>> from the Johns Hopkins Bloomberg School of Public Health and would like to talk to you about our research study on the effects of adding a cooking skills intervention to the Diabetes Prevention Program.

- We are interested in how participating in such an intervention can impact weight loss, diet and food related knowledge.
- We ask you to join our study because you have not participated in the DPP before, but are eligible to do so. You do not have to join, it is your choice. There will be no penalty if you decide not to join. You can still do the DPP even if you choose not to participate in the research study.
- If you say yes, we will ask you to do a few things. First, we will ask you to give us permission for your DPP lifestyle coach to share your weight data with us that they collect every week.
- There will be two kinds of DPP groups. One groups will have regular DPP. The other group will have regular DPP plus 6 cooking classes throughout the first 4 months of the DPP. Each class will take 2 hours. Whether or not you are in the regular DPP group or the DPP group that also has cooking classes will be decided by random chance before the DPP starts.
- DPP classes will be virtual over Zoom. Cooking classes will be in person if COVID rates
  are low. If not, cooking classes will be virtual over Zoom and we will deliver food for
  you to cook to your home.
- Whichever DPP group you are in we will ask you to answer a few online surveys at the start of the study, after 4 months, and again at the end of the study. The surveys should take about an hour total each time.
- We will ask you to take pictures of everything you eat for 3 days at the start of the study. We will ask you to do this again for another 3 days at 4 months into the study. You will use an app on your phone called SmartIntake to do this, and we will help you remember to take photos and help you learn how to use the app. If you are familiar with MyFitnessPal, this is a similar way to track what you eat. Finally, we will also invite you to share your thoughts with us about the DPP program and the cooking classes at the end of the study.
- This study does not present any risks to you beyond those of daily living. All survey data collection will take place in your home, at your convenience. It is possible that you may injure yourself while you are cooking during the hands-on cooking classes, but that risk is



no more than it would be in everyday life. There may also be risk of food allergy events during the cooking classes, but again, this risk is no higher than in daily life. To avoid food allergy events, prior to any food tasting or cooking activities we will ask participants about any known food allergies, and will clearly identify all ingredients in the recipes we prepare and taste. As with all data collection, there is the possibility of breach of confidentiality.

- To protect your confidentiality, we will not collect any sensitive information. Moreover, any information that we do collect will be immediately de-identified and only participant ID codes will be used on all quantitative and qualitative data. We will need to contact you by phone and email. We may need to collect your address so we can deliver food to you for virtual cooking classes. But we will not collect any other identifying information about you. Your name will never be published and will be kept confidential.
- There is a risk that someone outside the study will see your information. We will do our best to keep your information safe by using a special code to identify you. We will also keep your information separate, and will keep all data on locked computers and secure servers. We will delete all identifying information when your participation is complete. Any transcripts from interviews or photographs will be linked to an anonymous ID number, not to your name.
- Through your participation in this study you may learn new skills related to cooking and food agency. You may also develop insights into your cooking and food choices that may lead to making positive health changes. Attending cooking classes focused on diabetes prevention and documenting your meals may also lead you to think in new ways about how you prepare food as well. We hope this knowledge will help ourselves and others design better cooking classes for other DPP participants.
- We will let the community know about the results of the study. Results will likely be published but your name will never be used.
- You will receive a \$100 total as compensation for your completed participation in the research study. You will receive \$20 after the first round of data collection, \$20 after the data collection at 4 months, and \$60 after the 12-month data collection.
- If you are in the cooking class group you will also get food during the cooking classes and a recipe book to keep. If you are in the regular DPP group, you will get the recipe book and the opportunity to take a cooking class after data collection for the study ends.
- Your study information is protected by a Certificate of Confidentiality. This Certificate allows us, in some cases, to refuse to give out your information even if requested using legal means.
- It does not protect information that we have to report by law, such as child abuse or some infectious diseases. The Certificate does not prevent us from disclosing your information if we learn of possible harm to yourself or others, or if you need medical help.
- Disclosures that you make yourself about your study information are not protected.



- Do you have any questions? [Probe to assess the participant's understanding.]
- Would you like to join the study?
- You may contact Dr. Julia Wolfson about your questions or problems with this work.
- Call or contact the **Johns Hopkins Bloomberg School of Public Health IRB Office** if you have questions about your rights as a study participant. Contact the IRB if you feel you have not been treated fairly or if you have other concerns. The IRB contact information is:

Telephone: 410-955-3193 Toll Free: 1-888-262-3242 E-mail: jhsph.irboffice@jhu.edu

- [If yes] Thank you. We will be in contact to schedule the next steps.
- [If no] Thank you for your time. We understand and we wish you the best.